CLINICAL TRIAL: NCT03039738
Title: A Prospective Evaluation of Surveillance Monitoring as an Alternative to Telemetry in Patients Scheduled for Telemetry Without American Heart Association (AHA) Indication
Brief Title: Surveillance Monitoring as an Alternative to Telemetry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medtronic shift in strategic direction for study device
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COVMOPO0561
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-04

CONDITIONS: Telemetry; Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Telemetry Monitoring Arm (Active Comparator): The telemetry group will serve as the control group and will be monitored via the site's standard of care telemetry protocols.
  Interventions: Device: Telemetry Monitoring
- Surveillance Monitoring Arm (Experimental): Subjects in the surveillance monitoring group will alternatively be admitted to medical surgical unit and be monitored via the surveillance monitoring platform.
  Interventions: Device: Vital Sync IM & VPMP (Surveillance Monitoring)

INTERVENTIONS:
Device: Vital Sync IM & VPMP (Surveillance Monitoring) — The Vital Sync™ Informatics Manager (IM) & Virtual Patient Monitoring Platform (VPMP) is an electronic medical record connectivity and remote continuous patient monitoring software solution.
  Arms: Surveillance Monitoring Arm
Device: Telemetry Monitoring — Continuous ECG monitoring for hospitalized patients at-risk for cardiac events.
  Arms: Telemetry Monitoring Arm

SUMMARY:
The purpose of the study is to evaluate the impact of surveillance monitoring versus telemetry monitoring on clinical, healthcare economics, resource utilization, and qualitative outcomes.

DETAILED DESCRIPTION:
This will be single-center, prospective, pilot, pre/post implementation study to collect post-market data on hospitalized subjects monitored via telemetry and surveillance monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent by subject
2. Male or female 18 years of age or older
3. Expected hospitalized admission on the general care floor or medical surgical unit for at least one overnight stay and/or > 12 hours
4. Scheduled for telemetry monitoring
5. Diagnosis indicates American Heart Association (AHA) telemetry Class III or none and therefore not indicated for telemetry monitoring
6. For surveillance monitoring group subjects, treating provider who scheduled subject for telemetry agrees to alternative monitoring plan of surveillance monitoring
7. Willingness to have study devices attached and hair shaved at sensor location as needed during study participation
8. Willingness to participate in all aspects of the study

Exclusion Criteria:

1. Implanted pacemaker or atrial defibrillator
2. Allergy or sensitivity to ECG leads or adhesives that are similar to ECG leads
3. Current AHA Class I or II indication/prescription for telemetry monitoring
4. Prescription for other continuous condition monitoring such as capnography or pulse oximetry
5. Ongoing opioid therapy by patient-controlled analgesia (PCA), by epidural or intrathecal infusions or by intravenous analgesia, per Investigator discretion
6. Ventilated or intubated patients at the time of enrollment
7. Female subject is pregnant, lactating, trying to get pregnant, or has a positive pregnancy test for women with childbearing potential
8. Condition that, in the opinion of the investigator, may prevent completion of the study or protocol requirements
9. Subject is considered as being morbidly obese (defined as BMI >50.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey House, MD, PhD, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telemetry Monitoring Arm | Surveillance Monitoring Arm
Started | 206 | 0 (This arm did not initiate. The study was terminated following the completion of the telemetry phase.)
Completed | 152 | 0
Not Completed | 54 | 0
Not completed — Incomplete data sets | 54 | 0

BASELINE CHARACTERISTICS:
Population: The Surveillance Monitoring Arm did not initiate as the study was terminated following the completion of the TM phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemetry Monitoring Arm | Surveillance Monitoring Arm | Total
Number analyzed (Participants) | 206 | 0 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (15.6) |  | 55.3 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 |  | 107
  Male | 99 |  | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 |  | 3
  Not Hispanic or Latino | 202 |  | 202
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 152 |  | 134
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (9.2) |  | 28.8 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay (LOS) as Assessed by Review of Medical Records
Description: LOS will be determined by comparing LOS Between the Surveillance Monitoring and Telemetry Monitoring Period Arms.
Time Frame: Baseline to end of hospital stay (or up to 30 day post enrollment)
Population: The study was prematurely terminated; no conclusion should be drawn from the reported data. Data for SM arm were not collected.
Measure: Mean (Standard Deviation); unit: hrs
Groups:
- Telemetry Monitoring (TM) Arm: The telemetry group will serve as the control group and will be monitored via the site's standard of care telemetry protocols.
  Telemetry Monitoring: Continuous ECG monitoring for hospitalized patients at-risk for cardiac events.
- Surveillance Monitoring (SM) Arm: Subjects in the surveillance monitoring group will alternatively be admitted to medical surgical unit and be monitored via the surveillance monitoring platform.
  Vital Sync IM & VPMP (Surveillance Monitoring): The Vital Sync™ Informatics Manager (IM) & Virtual Patient Monitoring Platform (VPMP) is an electronic medical record connectivity and remote continuous patient monitoring software solution.
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 152 | 0
hrs | 79.9 (73.0) |

2. Secondary Outcome: Associated Health Care Costs (HCC) as Determined by Review of Billing Records
Description: Health Care Costs will be determined by comparing HCC between the surveillance monitoring and telemetry monitoring arms
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: The study was prematurely terminated; the billing data for both TM and SM arms were not collected, and outcome measure analysis was not performed.
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Hospital Unit Transfers (HUT) as Determined by Review of Medical Records
Description: Hospital Unit Transfers (HUT) will be determined by comparing the number of hospital unit transfers between monitoring arms.
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: The study was prematurely terminated; the data for SM Arm were not collected, and no outcome measure analyses were performed. No conclusion should be drawn from the reported data.
Measure: Count of Participants; unit: Participants
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 152 | 0
Participants | 143 |

4. Secondary Outcome: Length of Stay (LOS) in the ICU as Determined by Review of Medical Records
Description: Length of Stay in the ICU will be determined by comparing numbers between monitoring arms.
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: The study was prematurely terminated; the data for SM Arm were not collected, and no outcome measure analyses were performed. No conclusion should be drawn from the reported data. Only participants who were admitted to ICU, were assessed for this Outcome.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 5 | 0
hrs | 4.4 (4.9) |

5. Secondary Outcome: Number of Participants With Clinical Interventions (CI) as Determined by Review of Medical Records
Description: CI include Rapid Response Team calls and Code Blue Activations. The Number of Clinical Interventions will be determined by comparing numbers between monitoring arms.
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 152 | 0
Participants | 14 |

6. Secondary Outcome: Time of Rapid Response Team Activation to Time of a Threshold Notification as Measured by the Surveillance Monitoring System Only
Description: Time of Rapid Response Team (RRT) will be determined by comparing the number of RRT interventions between monitoring arms (only for surveillance monitoring arm)
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: The study was prematurely terminated; this outcome was for Surveillance Monitoring arm only. The data were not collected, and no outcome measure analysis was performed.
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Clinical Team and Patient Satisfaction as Measured by Qualitative Questionnaires
Description: Clinical Team and Patient Satisfaction will be determined by comparing the Qualitative Questionnaire response between monitoring arms.
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: The patient and clinical team satisfaction questionnaires were designed to be collected for the SM arm only. The study enrolled control arm only prior to termination. The questionnaires were not collected, and no outcome measure analyses were performed.
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Clinicians Familiarity With AHA Guidelines and Telemetry Utilization as Measured by Qualitative Questionnaires
Description: Number of clinicians "very familiar" and "somewhat familiar" with AHA guidelines was reported. The questionnaire was administered to all clinicians (e.g. ED physicians, nurses, critical care nurses, intensivists, and hospitalists) involved in the care of study participants at each hospital; it was not administered to study subjects.
Time Frame: Baseline to end of hospital stay (or up to 30 days post enrollment)
Population: All clinicians (e.g. ED physicians, nurses, critical care nurses) involved in the care of study participants at each hospital (not study subjects.) The study was prematurely terminated; no conclusion should be drawn from the reported data. The data for SM Arm were not collected, and no outcome measure analyses were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Telemetry Monitoring (TM) Arm | Surveillance Monitoring (SM) Arm
Number analyzed (Participants) | 259 | 0
Participants | 118 |

ADVERSE EVENTS:
Time Frame: The recording of adverse events for all enrolled subjects began after the telemetry devices were attached and ended with the subject completing study enrollment. Completion is defined by when a subject is discharged from the hospital, completes 30 day (± 2 days) enrollment period, or if the subject is withdrawn from the study for any reason.
Description: Only the following adverse events were collected for this study:
  * Any adverse events noting mild or moderate physiological deterioration
  * Any adverse event whose relationship to the study device is: possible, probable, definite, or unknown/ impossible to determine, regardless of what the event may be.
  * All serious adverse event, of any relationship, meeting the protocol definitio
Arm/Group | Telemetry Monitoring Arm | Surveillance Monitoring Arm
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/0
Serious Adverse Events (participants affected / at risk) | 40/206 | 0/0
Other Adverse Events (participants affected / at risk) | 8/206 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telemetry Monitoring Arm (N=206) | Surveillance Monitoring Arm (N=0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | NA
AGITATED DELIRIUM (Psychiatric disorders) | 1 | NA
ALTERED MENTAL STATUS (Psychiatric disorders) | 2 | NA
APHASIA (Nervous system disorders) | 1 | NA
ASPIRATION PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | NA
CARDIAC ARREST (Cardiac disorders) | 2 | NA
EXPRESSIVE APHASIA (Nervous system disorders) | 1 | NA
FACIAL EDEMA (CONCERN FOR ALLERGIC REACTION VS. ATYPICAL ANGIOEDEMA) (General disorders) | 1 | NA
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 | NA
GROSS HEMATURIA (Renal and urinary disorders) | 1 | NA
HEMORRHAGIC SHOCK (GI BLEED SOURCE) (Vascular disorders) | 1 | NA
HYPERCAPNIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | NA
HYPERCARBIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | NA
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 | NA
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 | NA
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | NA
HYPOTENSION (Vascular disorders) | 3 | NA
HYPOXEMIA (Respiratory, thoracic and mediastinal disorders) | 1 | NA
LETHARGY (Nervous system disorders) | 1 | NA
NEW ONSET ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RESPONSE (Cardiac disorders) | 1 | NA
NEW ONSET ATRIAL FIBRILLATION/FLUTTER (Cardiac disorders) | 1 | NA
NON ST ELEVATION MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | NA
NON STEMI (Cardiac disorders) | 3 | NA
NON SUSTAINED VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 | NA
RECURRENT HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | NA
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | NA
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | NA
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | NA
SYMPTOMATIC BRADYCARDIA (Cardiac disorders) | 1 | NA
TRANSFUSION-INDUCED PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | NA
UNRESPONSIVENESS/HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | NA
UNRESPONSIVENESS/RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | NA
WORSENING ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | NA
WORSENING ANEMIA (Blood and lymphatic system disorders) | 4 | NA
WORSENING AV FISTULA INFECTION (Infections and infestations) | 1 | NA
WORSENING CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 | NA
WORSENING COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 | NA
WORSENING DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | NA
WORSENING GASTROINTESTINAL BLEED (Gastrointestinal disorders) | 2 | NA
WORSENING HYERKALEMIA (Metabolism and nutrition disorders) | 1 | NA
WORSENING HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 | NA
WORSENING HYPERKALEMIA (Metabolism and nutrition disorders) | 3 | NA
WORSENING HYPERTENSION (Vascular disorders) | 4 | NA
WORSENING HYPOKALEMIA (Metabolism and nutrition disorders) | 2 | NA
WORSENING HYPONATREMIA (Metabolism and nutrition disorders) | 1 | NA
WORSENING HYPOTENSION (Vascular disorders) | 2 | NA
WORSENING METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | NA
WORSENING QT PROLONGATION (Investigations) | 1 | NA
WORSENING SEVERE SEPSIS (Infections and infestations) | 1 | NA
WORSENING SINUS BRADYCARDIA (Cardiac disorders) | 1 | NA
WORSENING SINUS TACHYCARDIA (Cardiac disorders) | 1 | NA
WORSENING TACHYCARDIA (Cardiac disorders) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telemetry Monitoring Arm (N=206) | Surveillance Monitoring Arm (N=0)
AGITATION (Psychiatric disorders) | 1 | NA
CHEST PAIN (General disorders) | 2 | NA
HYPOTENSION (Vascular disorders) | 1 | NA
INCREASED ALTERED MENTAL STATUS (Psychiatric disorders) | 1 | NA
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | NA
WORSENING LETHARGY (Nervous system disorders) | 1 | NA

LIMITATIONS AND CAVEATS:
This study was terminated early, no conclusions should be drawn from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03039738/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT03039738/SAP_001.pdf